CLINICAL TRIAL: NCT05659485
Title: Measuring Family Engagement in Care (The FAME Study)
Acronym: FAME
Status: Recruiting | Type: Observational
Sponsor: Lady Davis Institute (Other)
Collaborators: Jewish General Hospital (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Michael Goldfarb, Attending Staff, Division of Cardiology, Lady Davis Institute
Other Study IDs: 2022-3191
Record Dates: First submitted 2022-12-05; First posted 2022-12-21 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Family Engagement; Patient-centered Care; Critical Care
Keywords: Family; Engagement; Family engagement; Family-centered care; Measures; Instruments; Intensive care unit

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
There are currently no validated tools to specifically measure family engagement in the intensive care unit (ICU). To address this gap, an interdisciplinary team developed a novel instrument to measure family engagement in the ICU. This will be a prospective observational cohort with an embedded qualitative study to validate the FAMily Engagement (FAME) instrument in the ICU setting. This study will also evaluate the association between family activation, engagement, and family-centred outcomes, and exploring factors (age, relationship, sex, gender, race/ethnicity) that may influence family engagement in the ICU.

DETAILED DESCRIPTION:
This will be a prospective observational cohort study of 198 family members in the ICUs of 4 Canadian hospitals in 3 provinces (Alberta, Ontario, and Quebec) over a 12-week period. These sites were chosen due to their urban setting and distant geographic range to capture differing practice patterns, a higher percentage of racialized patients, and language and cultural differences. The target recruitment is 50 family members from each participating site. A "family member" will be considered anyone with a biological, legal, or emotional relationship with the patient and whom the patient would want involved in their care.

ELIGIBILITY:
Inclusion Criteria:

* Family member of patient admitted to the intensive care units
* Able to participate in English or French
* Age 18 years old or older

Exclusion Criteria:

* ICU stays less than 24 hours
* Another family member has already participated in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Family members, aged 18 years old or older, of patients admitted to intensive care units. The term "Family member" includes anyone that has a biological, legal, or emotional relationship with the patient and the patient would like to be involved in their care.
Sampling Method: Non-Probability Sample
Enrollment: 198 (Estimated)
Dates: Start 2023-01-31 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Family engagement in care (as measured by FAME) | Within 24 hours of enrolment
  The FAMily Engagement (FAME) questionnaire is an instrument developed to assess current family engagement practice. Items address key principles of family-centered care, such as dignity and respect, information sharing, participation, and collaboration. They also address family engagement domains, including family presence, family needs, communication and education, decision making, and direct care. A five-point Likert scale (1=strongly agree, 2=agree, 3=neutral, 4=disagree, 5=strongly disagree) is used for responses, which are then transformed to a 0-100 scoring system, with higher scores indicating greater engagement in care and lower scores indicating lesser engagement in care. The overall engagement score is calculated by dividing the sum of the scores by the number of questions answered, with the result ranging from 0-100.

SECONDARY OUTCOMES:
Family activation (as measured by FAM-Activate) | Within 24 hours of enrolment
  FAM-Activate is a 4-question measure that assesses the family member's knowledge, skills, and confidence concerning care participation.
Family mental health (as measured by HADS) | Within 2 weeks of hospital discharge.
  The Hospital Anxiety and Depression Scale (HADS) survey is a validated self-reported instrument to measure anxiety and depression in medical patients. The survey consists of 14 questions (7 depression-related and 7 anxiety-related) which are scored on a 4-point Likert scale (0-3). The sum of the sub-scores on each of the two subscales (anxiety and depression) represents the total score. A lower total score indicates a milder condition whereas a higher total score indicates a higher level of distress.
Family care satisfaction (as measured by FS-ICU 24) | Within 2 weeks of hospital discharge.
  The Family Satisfaction in the ICU survey (FS-ICU 24) is a validated 24-item self-report instrument that assesses family satisfaction and experience with care in the ICU.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Goldfarb, MD MSc, Principal Investigator — Lady Davis Institute
Locations (6):
- Canada (6):
  - Foothills Medical Centre, Calgary, Alberta
  - St. Michael's Hospital, Toronto, Ontario
  - Jewish General Hospital / Lady Davis Institute, Montreal, Quebec
  - Centre hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec
  - Montreal General Hospital, Montreal, Quebec
  - Royal Victoria Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barello S, Castiglioni C, Bonanomi A, Graffigna G. The Caregiving Health Engagement Scale (CHE-s): development and initial validation of a new questionnaire for measuring family caregiver engagement in healthcare. BMC Public Health. 2019 Nov 27;19(1):1562. doi: 10.1186/s12889-019-7743-8. PMID 31771546
- [Background] Brown SM, Rozenblum R, Aboumatar H, Fagan MB, Milic M, Lee BS, Turner K, Frosch DL. Defining patient and family engagement in the intensive care unit. Am J Respir Crit Care Med. 2015 Feb 1;191(3):358-60. doi: 10.1164/rccm.201410-1936LE. No abstract available. PMID 25635496
- [Background] Anderson WG, Arnold RM, Angus DC, Bryce CL. Posttraumatic stress and complicated grief in family members of patients in the intensive care unit. J Gen Intern Med. 2008 Nov;23(11):1871-6. doi: 10.1007/s11606-008-0770-2. Epub 2008 Sep 9. PMID 18780129
- [Background] Devlin JW, Skrobik Y, Gelinas C, Needham DM, Slooter AJC, Pandharipande PP, Watson PL, Weinhouse GL, Nunnally ME, Rochwerg B, Balas MC, van den Boogaard M, Bosma KJ, Brummel NE, Chanques G, Denehy L, Drouot X, Fraser GL, Harris JE, Joffe AM, Kho ME, Kress JP, Lanphere JA, McKinley S, Neufeld KJ, Pisani MA, Payen JF, Pun BT, Puntillo KA, Riker RR, Robinson BRH, Shehabi Y, Szumita PM, Winkelman C, Centofanti JE, Price C, Nikayin S, Misak CJ, Flood PD, Kiedrowski K, Alhazzani W. Clinical Practice Guidelines for the Prevention and Management of Pain, Agitation/Sedation, Delirium, Immobility, and Sleep Disruption in Adult Patients in the ICU. Crit Care Med. 2018 Sep;46(9):e825-e873. doi: 10.1097/CCM.0000000000003299. PMID 30113379
- [Background] Goldfarb M, Bibas L, Burns K. Patient and Family Engagement in Care in the Cardiac Intensive Care Unit. Can J Cardiol. 2020 Jul;36(7):1032-1040. doi: 10.1016/j.cjca.2020.03.037. Epub 2020 Mar 31. PMID 32533931
- [Background] Goldfarb MJ, Bechtel C, Capers Q 4th, de Velasco A, Dodson JA, Jackson JL, Kitko L, Pina IL, Rayner-Hartley E, Wenger NK, Gulati M; American Heart Association Council on Clinical Cardiology; Council on Cardiovascular and Stroke Nursing; Council on Lifelong Congenital Heart Disease and Heart Health in the Young; Council on Cardiovascular Radiology and Intervention; Council on Hypertension; Council on the Kidney in Cardiovascular Disease; and Council on Lifestyle and Cardiometabolic Health. Engaging Families in Adult Cardiovascular Care: A Scientific Statement From the American Heart Association. J Am Heart Assoc. 2022 May 17;11(10):e025859. doi: 10.1161/JAHA.122.025859. Epub 2022 Apr 21. PMID 35446109
- [Background] Goldfarb MJ, Bibas L, Bartlett V, Jones H, Khan N. Outcomes of Patient- and Family-Centered Care Interventions in the ICU: A Systematic Review and Meta-Analysis. Crit Care Med. 2017 Oct;45(10):1751-1761. doi: 10.1097/CCM.0000000000002624. PMID 28749855
- [Background] Goldfarb M, Debigare S, Foster N, Soboleva N, Desrochers F, Craigie L, Burns KEA. Development of a Family Engagement Measure for the Intensive Care Unit. CJC Open. 2022 Aug 5;4(11):1006-1011. doi: 10.1016/j.cjco.2022.07.015. eCollection 2022 Nov. PMID 36444373
- [Derived] Duong J, Kifell J, Gelinas C, Udupa S, Beydoun SA, Stephenson A, Goldfarb M. Validation of the French-Canadian Version of FAME, a Family Engagement Measurement Tool for the Intensive Care Unit. Can J Nurs Res. 2026 Mar;58(1):78-85. doi: 10.1177/08445621251385620. Epub 2025 Oct 15. PMID 41091932